CLINICAL TRIAL: NCT01524939
Title: Multicenter, Single-arm, Phase IV Study to Evaluate the Efficacy, Safety of Combined Therapy of Aspirin and High Dose "IVIG-SN" in Pediatric Patients With Kawasaki Disease
Brief Title: Study of Combined Therapy of Aspirin and "IVIG-SN" in Kawasaki Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVIG-SN_KD_P4
Record Dates: First submitted 2012-01-25; First posted 2012-02-02 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-01

CONDITIONS: Kawasaki Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational product (Experimental)
  Interventions: Drug: immunoglobulin G

INTERVENTIONS:
Drug: immunoglobulin G — Intravenously administer a single dose of the product (2g/kg) for at least 12 hours

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and of Immune Globulin Intravenous (Human) IVIG-SN™ in subjects with kawasaki diseases.

DETAILED DESCRIPTION:
This clinical trial was designed as a multicenter, single-arm, and open-label clinical trial.

Evaluate the incidence of coronary artery lesions in the 7th week of IVIG-SN administration, compared to the incidence of coronary artery lesions among untreated Kawasaki patients, to prove the superior efficacy of IVIG-SN.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients aged 6 months - 5 years
2. Case definition for complete KD: Fever (≥ 38.5°C) for ≥ 5 days (but less than 10 days), 4/5 standard clinical criteria
3. Case definition for incomplete KD: Fever ≥ 5 days(but less than 10 days) and 3 clinical criteria plus coronary artery lesion on echocardiogram.
4. Subjects whose parents or legally acceptable representative (LAR) gave voluntary written consent to participate in this clinical trial

Exclusion Criteria:

1. Those whose blood test results show abnormalities of significance as follows : Platelet count < 100,000/mm3, WBC count <3,000 cells/mm3,Those whose hemogloblin, hematocrit or red blood cell count exceed 30% of the upper limit of the normal range or are 30% below the lower limit of the normal range.
2. Those who have been administered other clinical product in the last 30 days after this clinical trial commenced
3. Those who have been administered TNF alpha or steroid within 48 hours after being administered the test product
4. Those who plan to be inoculated with live vaccine during the clincial trial period
5. Those considered difficult to participate in clinical trial due to serious chronic diseases(e.g., cardiovascular diseases except controllable hypertension, diseases of the respiratory system concurrent with respiratory failure, metabolic disease, kidney dysfunction, hemoglobinopathy, etc.)
6. Those who have been administered an immunosuppressant or immune modifying drug in the last 3 months before the innoculation with the test product
7. Those who are HIV-positive or have immune dysfunctions including immunodeficiency
8. Those who have previously exhibited hypersensitivity or shock to IVIG agents
9. Patients with underlying liver disease or liver dysfunction with known etiology.
10. Patients with kidney dysfunction, whose Creatinine level is found to be over 2 times higher than the upper limit of the normal ranges in a screening test
11. Those who have -- or previously had -- a malignant tumor
12. Those who have previously been diagnosed with IgA deficiency
13. Those found unsuitable for undergoing the tests

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Incidence of coronary artery lesions | 7 weeks
  Incidence of coronary artery lesions in the 7 weeks after IVIG-SN infusion

SECONDARY OUTCOMES:
Incidence of coronary artery lesions | 2weeks
  Incidence of coronary artery lesions in the 2nd week after IVIG-SN infusion
Total fever duration | baseline
  Total fever duration after IVIG-SN infusion
variation of ESR, CRP, NT-proBNP,CK-MB | baseline
  Evaluation in variation of ESR, CRP, NT-proBNP or BNP, and CK-MB

CONTACTS AND LOCATIONS:
Overall Officials: June Huh, MD,Ph.D, Principal Investigator — Samsung Medical Center
Locations (7):
- South Korea (7):
  - Wonju christian Hospital, Wŏnju, Kang-won
  - Gachon University Gil Hospital, Incheon
  - Asan Medical center, Seoul
  - Kyung Hee university at Gangdong, Seoul
  - Kyung Hee university medical center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul ST. Mary's Hospital, Seoul